CLINICAL TRIAL: NCT04294875
Title: Phase l, First in Human, Multi-centre, Open-label, Clinical Trial of MPT0B640 in Subject With Locally Advanced or Metastatic Solid Malignancies
Brief Title: Phase I, FIH, MTD for MPT0B640, Multi-centre, Open-label, Subject With Locally Advanced or Metastatic Solid Malignancies
Acronym: MPT0B64
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study held.
Sponsor: J Ints Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JO201901-01
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MPT0B640 (Other): There is Single Arm in this Clinical Trials.
  Interventions: Drug: MPT0B640

INTERVENTIONS:
Drug: MPT0B640 — PO, every 3 days. dose escalation per MTD

SUMMARY:
Phase l, First in Human, Multi-centre, Open-label, Clinical Trial of MPT0B640 in Subject with Locally Advanced or Metastatic Solid Malignancies

Phase I. Advanced or metastatic solid malignancy First in Human. HSP90 inhibitor Multi-center clinical trials. Open label.

To determine the maximum tolerated dose (MTD) or maximum feasible dose (MFD) of MPT0B640

DETAILED DESCRIPTION:
Classical 3+3 design to determine the maximum tolerated dose (MTD) or maximum feasible dose (MFD) of MPT0B640 .

Up to 9 times of administration, Oral suspension, once every 3rd day.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all inclusion criteria as listed below:

1. Histologically or cytologically confirmed, locally advanced or metastatic solid malignancies, such as non-small cell lung cancer (NSCLC), breast cancer, hepatocellular carcinoma, colorectal, prostate and pancreatic cancer who is not suitable for surgery or radiotherapy.
2. Subjects who have progressed after receiving all available standard treatment known to confer clinical benefit or for which no effective therapy exists.
3. Radiological documentation of disease progression while on a previous treatment.
4. Discontinued all previous treatment for cancer for at least 14 days and recovered from the effects of therapy.
5. Eastern Cooperative Oncology Group (ECOG) 0 ~ 1
6. 19 years and older of age (Adult)
7. At least one measurable lesion by Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
8. Laboratory values: Hematologic parameters must be met without recent transfusions within 7 days of enrolment.

   1. Serum creatinine < 1.5× upper limit of normal (ULN) or if higher than normal range, calculated creatinine clearance (CrCl) must be ≥ 60mL/min/1.73m2 (by Cockroft-Gault formula); actual body weight must be used for CrCl unless body mass index (BMI) > 30kg/m2 then lean body weight must be used
   2. Total bilirubin ≤ 1.5×ULN (except for Gilbert's syndrome which will allow bilirubin ≤2.0 ×ULN).
   3. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5×ULN, or ≤ 5×ULN if due to liver involvement by tumour.
   4. Haemoglobin ≥ 9.0g/dL.
   5. Platelets ≥ 100×109cells/L.
   6. Absolute neutrophil count ≥ 1.5×109cells/L.
9. Subjects signed informed contents form
10. Expected lifespan ≥ 3 months
11. Female should be using adequate contraceptive measures, e.g., use at least two of the following types of appropriate and effective birth control from 2 weeks prior to the first dose of the study drug until 90 days after last dose. One of these methods must be a double barrier method (condom with diaphragm plus spermicidal agent [foam/gel/cream/film/suppository]). Additional methods are IUD or IUS, vasectomy by sole male partner and use of approved oral, injected, or implanted hormonal methods of contraception.
12. Female should not breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential at screening.
13. Male subjects should be willing to use barrier contraception include using one of the following during the study and for 90 days after last dose of the study drug. (Abstinence, condom plus spermicidal agents [foam gel/cream/film/suppository])

Exclusion Criteria Any subject meeting one or more of the following exclusion criteria may not be entered into the trial.

1. Symptomatic central nervous system (CNS) metastases which are neurologically unstable or requiring increasing doses of steroids within the 28 days prior to study entry to control their CNS disease and require local CNS-directed therapy
2. Systemic anticancer treatment 14 days prior to the first dose of study drug on Visit 1
3. Subjects who have undergone any major surgery* (as judged by the investigator, excluding placement of vascular access) ≤ 28 days of the first dose of study drug on Visit 1 or who have not recovered from side effects of such therapy

   *Major surgery defined as a surgical operation within or upon the contents of the abdominal, pelvic, cranial or thoracic cavities and a procedure which given the locality, condition of patient, level of difficulty or length of time to perform, constitutes a hazard to life or function of an organ or tissue. Major surgery usually requires general anesthesia, a period of hospitalization of varying length (often a week) and may be performed by a surgical subspecialist.
4. Limited-field radiotherapy ≤ 7 days or extended-field thoracic radiotherapy < 28 days of study drug on Visit 1
5. Subjects with

   1. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 480 milliseconds (ms) (CTCAE grade 1) using Frederica's QT correction formula.
   2. A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
   3. The use of concomitant medications that prolong the QT/QTc interval.
6. Subjects with impaired cardiac function or clinically significant cardiac disease such as:

   1. Left ventricular ejection fraction < 50%.
   2. Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA Grade ≥ 2), uncontrolled hypertension, or clinically significant arrhythmia.
   3. History of acute myocardial infarction or unstable angina pectoris < 6 months prior to study entry.
7. Subjects who had a prior history of another malignancy over the last 5 years
8. Subjects able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major restriction of the stomach or bowels
9. Subjects with active human immunodeficiency virus (HIV) or hepatitis B or C infection
10. Subjects who were administered another investigational product within 3 weeks prior to screening
11. Subjects with any unresolved toxicity of Grade ≥ 2 from previous anti-cancer treatment, except for alopecia and skin pigmentation.
12. Subjects with any clinically significant abnormal intestinal findings that may interfere with the administration, passage, or absorption of the investigational product, which makes the subjects unable to orally take the suspension form of drugs.
13. Subjects with drug abuse and unstable medical, psychological or social conditions that may interfere with participating in the study or assessment of the results of the study
14. Subjects with any condition or illness might compromise subject safety or interfere with the evaluation of the safety of the drug by investigator's decision
15. Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry
16. According to investigator's judgement, protocols cannot be followed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
MTD of the dose of MPT0B640 | 28days(+/-2days)

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Seah, Study Director — J Ints Bio